CLINICAL TRIAL: NCT01176110
Title: A Randomized Pilot Study for Thermal Management in Patients With Interventional Minimally Invasive Valve Replacement
Brief Title: Thermal Management in Patients With Interventional Minimally Invasive Valve Replacement
Acronym: TIMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: PD Dr. Michael Sander, Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum Charité - Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TIMI101; EA1/142/10 (Other: ethics commitee)
Record Dates: First submitted 2010-07-29; First posted 2010-08-05 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-07

CONDITIONS: Outcomes; Body Temperature
Keywords: hypothermia; minimal invasive valve replacement
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thermal management with LMA PerfecTemp™ (Experimental)
  Interventions: Device: LMA Perfect Temp
- no specific thermal management (Active Comparator)
  Interventions: Device: LMA Perfect Temp

INTERVENTIONS:
Device: LMA Perfect Temp — The LMA PerfecTemp™ patient warming system combines warming beneath the patient and advanced pressure reduction to combat hypothermia and decubitus ulcers. This device is used during the interventional minimal invasive valve replacement with unprecedented ease and safety

SUMMARY:
It is known that perioperative hypothermia can influence the postoperative outcome negatively.

The most important complications are cardiac, increased blood loss with need for transfusion and a significantly increased wound infection rate.

The thermal redistribution after the induction of anesthesia is on of the reasons for perioperative hypothermia. Another reason is negative heat balance during surgery.

Further negative side effects of hypothermia are an increase of blood viscosity and thus a higher risk for thrombosis, coagulopathy and thus an increased risk of bleeding.

The aim of the study is to evaluate if patients with a perioperative active thermal management during an interventional minimal invasive valve replacement have a significantly higher body temperature at the end of the operation than patients without an active thermal management. Secondary outcome variables are complication rates, length of mechanical ventilation and length of ICU treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who need an interventional minimal invasive valve replacement
* Age ≥ 18 years
* scheduled general anesthesia during intervention
* no participation on another interventional study
* signed informed consent

Exclusion Criteria:

* pregnant or breast feeding women
* non-elective intervention
* conversion to HLM
* implantation of IABP
* pre-existing decubitus
* patients who are not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Temperature at the end of the intervention | average 2 hours
  The end of the surgical procedure is defined and is recorded for all patients in the hospital information systems. This time point will be used to record the body temperature at the end of the intervention

SECONDARY OUTCOMES:
hospital stay | max 28 days
mechanical ventilation time | maximum 28 days
  The mechanical ventilation time in the hospital is recorded electronically. The time frame will be recorded as the outcome measure in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, MD, Principal Investigator — Dept. of Anesthesiology Charité Universitaetsmedizin Berlin; Claudia Spies, MD, Study Chair — Dept. of Anesthesiology Charité Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Berlin, State of Berlin, Germany